CLINICAL TRIAL: NCT01132534
Title: A Randomized Study Comparing Endoscopic Video-Autofluorescence Imaging Followed by Narrow Band Imaging With Standard Videoendoscopy for the Detection of High Risk Lesions of Stomach
Brief Title: A Randomized Study Comparing Autofluorescence Imaging(AFI) Followed by Narrow Band Imaging(NBI) With Videoendoscopy for the Detection of High Risk Lesions of Stomach
Acronym: CAFBI
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: A/Prof Jimmy So, National University Hospital, Singapore
Other Study IDs: DSRB D/07/163
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-05

CONDITIONS: Gastric Cancer
Keywords: OGD; NBI; AFI; Videoendoscopy; Narrow Band Imaging; Autofluorescence Imaging
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SE then AFI/NBI: Patients will be randomised to be examined by standard videoendoscopy (SE) then combined AFI/NBI during the esophagogastroduodenoscopy (EGD) examination at same setting.
- AFI/NBI then SE: Patients will be randomised to be examined by combined AFI/NBI then standard videoendoscopy (SE) during the EGD examination at same setting.

SUMMARY:
Videoendoscopy is the standard tool for examination of gastrointestinal tract. However, precancerous lesions and early gastric cancer can be easily missed by routine videoendoscopy. Autofluorescence Imaging (AFI) and Narrow band imaging (NBI) are 2 new imaging systems used in endoscopy which are recently developed. AFI based on the presence of natural tissue fluorescence on the gastrointestinal tract. By computation of the difference in the reflecting images, the system can reveal early cancers that are not detectable by standard endoscopy. NBI is a high resolution imaging using lights with narrowed wavelength range, which able to enhance the fine structure of the mucosa. Recent studies suggested combined AFI and NBI can improve the detection of early esophageal and gastric cancers.

The investigators are conducting a prospective randomized cross-over study to compare the accuracy between this combined AFI/NBI imaging with standard videoendoscopy in the detection of precancerous lesions and gastric cancer in a high risk population inSingapore. The investigators hypothesis is that this new combined imaging system improves the investigators detection of high risk lesions of stomach.

DETAILED DESCRIPTION:
Gastric cancer remains one of the leading causes of cancer deaths worldwide. Early detection and diagnosis of gastric cancer improves the outcomes of treatment. However, most of gastric cancers detected in Singapore are late and advanced in stages.

Videoendoscopy is the standard tool for examination of gastrointestinal tract. Despite the improvement of technology, early gastric cancers can be easily missed by routine examination, because there are few morphological changes. Therefore, a functional imaging modality, that can distinguish abnormal lesion from surrounding normal mucosa may complement the current videoendoscopy.

Autofluorescence Imaging (AFI) based on the presence of natural tissue fluorescence on the gastrointestinal tract. When the mucosa was exposed by an excitation light, certain endogenous molecules (fluorophores) will emit fluorescence light of longer wavelength. The fluorescent light can be detected and spectrally analyzed. By computation of the difference in the reflecting images, the system can specify lesions, including malignancies from the adjacent mucosa, and can reveal early cancers that are not detectable by standard endoscopy.

Narrow band imaging (NBI) is another novel optical imaging technique based on high resolution imaging, which aims at enhancing the fine structure of the mucosa. In NBI, the band widths of the red, blue, green components of the excitation light are narrowed to certain wavelength ranges, which allow better contrast of the superficial mucosa and the vascular structure. NBI has a maximum zoom capacity of 115 times. Abnormal lesions are detected by the presence of abnormal mucosal and vascular patterns.

Recent studies suggested that these AFI and NBI systems can be complementary to each other. The resolution of AFI is low but it can be used as a 'red flag' technique to screen any suspicious lesions from the normal mucosa. On the other hand, NBI produces high resolution images which allows detailed examination and subsequent target biopsy of the suspicious lesions based on AFI. Preliminary reports from Japan and the Netherlands suggested this combined imaging method improves the detection of early esophageal and gastric cancers. Recently, a new endoscopy system has been developed that incorporates standard videoendoscopy system with both AFI and NBI modes. By pressing a switch, the endoscopy system can switch from normal white light to either a narrow band light or autofluorescence mode. This novel system reduces the convenience and discomfort for the patients to avoid repeated intubation. The purpose of this study is to prospectively evaluate this combined imaging modality for detection of high risk gastric lesions and early cancers by comparing it with standard videoendoscopy in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=50
2. Ethnic Chinese
3. Presenting symptom - dyspepsia

Exclusion Criteria:

1. Patients who are unable to give an informed consent.
2. Patients with previous surgery of the stomach.
3. Patients presented with active gastrointestinal bleeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria of this study is based on our previous study "Dan YY, So JBY, Yeoh KG. Endoscopic screening for gastric cancer: Clin Gastroenterol Hepatol 2006;4:709-716." which showed that ethnic Chinese and aged 50 or above have increased risk of developing gastric cancer.
  In another study "Zhu F, Yeoh KG, So JBY, et al. Risk factors associated with intestinal metaplasia, a gastric pre-malignant lesion, in a chinese cohort under surveillance for gastric cancer: AACR; L.A. 2007 April" which is still ongoing, showed that the prevalence of intestinal metaplasia, a precancerous gastric lesion, is about 35% in this high risk population. Our sample size calculation is based on this finding and other relevant literature.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To compare the detection rate of premalignant lesions(intestinal metaplasia, gastric atrophy, dysplasia) and early neoplasia of stomach between combined AFI/NBI endoscopy versus standard endoscopy | 6 months
  The purpose of this study is to prospectively evaluate this combined imaging modality for detection of high risk gastric lesions and early cancers by comparing it with standard videoendoscopy in a randomized fashion.

SECONDARY OUTCOMES:
To assess the diagnostic accuracy AFI and NBI imaging | 6 months
  We aim to identify a method to improve our diagnosis of high risk gastric lesions in our population.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy BY So, MBChB, Principal Investigator — National University Hospital, Singapore

REFERENCES:
- [Derived] So J, Rajnakova A, Chan YH, Tay A, Shah N, Salto-Tellez M, Teh M, Uedo N. Endoscopic tri-modal imaging improves detection of gastric intestinal metaplasia among a high-risk patient population in Singapore. Dig Dis Sci. 2013 Dec;58(12):3566-75. doi: 10.1007/s10620-013-2843-2. Epub 2013 Sep 1. PMID 23996468